CLINICAL TRIAL: NCT02147132
Title: A Pilot Randomized, Placebo-Controlled, Crossover Study of the Effect of the Nicotine Nasal Spray and Varenicline on Cigarette Smoking Following Methadone Dosing in Methadone-Maintained Patients
Brief Title: Pilot Study of Nicotine Nasal Spray and Varenicline on Smoking in Methadone-Maintained Patients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Difficulty recruiting eligible participants; study medication was expiring.
Sponsor: University of Cincinnati (Other)
Responsible Party: Principal Investigator, Theresa Winhusen, Ph.D, University of Cincinnati
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2013-7275
Record Dates: First submitted 2014-05-19; First posted 2014-05-26 (Estimated); Results first posted 2018-12-05 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Cigarette Smoking; Methadone Maintenance
Keywords: Cigarette; Methadone; Smoking; Cessation; Varenicline; Nicotine
MeSH Terms: conditions — Cigarette Smoking; Smoking | interventions — Tobacco Use Cessation Devices; Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Order 1 (Experimental): Subjects assigned to this arm will receive Placebo Nasal Spray first (Week 1), followed by Nicotine Nasal Spray (Week 2), followed by Varenicline (Weeks 3-4), followed by a washout period (Week 5) and then Placebo Varenicline (Weeks 6-7).
  Interventions: Drug: Nicotine Nasal Spray; Drug: Varenicline; Drug: Placebo Nasal Spray; Drug: Placebo Varenicline
- Order 2 (Experimental): Subjects assigned to this arm will receive Placebo Nasal Spray first (Week 1), followed by Nicotine Nasal Spray (Week 2), followed by Placebo Varenicline (Weeks 3-4), followed by a washout period (Week 5) and then Varenicline (Weeks 6-7).
  Interventions: Drug: Nicotine Nasal Spray; Drug: Varenicline; Drug: Placebo Nasal Spray; Drug: Placebo Varenicline
- Order 3 (Experimental): Subjects assigned to this arm will receive Nicotine Nasal Spray first (Week 1), followed by Placebo Nasal Spray (Week 2), followed by Varenicline (Weeks 3-4), followed by a washout period (Week 5) and then Placebo Varenicline (Weeks 6-7).
  Interventions: Drug: Nicotine Nasal Spray; Drug: Varenicline; Drug: Placebo Nasal Spray; Drug: Placebo Varenicline
- Order 4 (Experimental): Subjects assigned to this arm will receive Nicotine Nasal Spray first (Week 1), followed by Placebo Nasal Spray (Week 2), followed by Placebo Varenicline (Weeks 3-4), followed by a washout period (Week 5) and then Varenicline (Weeks 6-7).
  Interventions: Drug: Nicotine Nasal Spray; Drug: Varenicline; Drug: Placebo Nasal Spray; Drug: Placebo Varenicline

INTERVENTIONS:
Drug: Nicotine Nasal Spray — 7 days. 1 mg/dose, up to 40x/day.
Drug: Varenicline — 14 days. Days 1-3: 0.5 mg once daily; Days 4-7: 0.5 mg twice daily; Days 8-14: 1 mg twice daily.
Drug: Placebo Nasal Spray — 7 days. 1 mg/dose, up to 40x/day.1 mg/dose, up to 40x/day. This will appear similar to the Nicotine Nasal Spray, but will be a placebo.
Drug: Placebo Varenicline — 14 days. Days 1-3: 0.5 mg once daily; Days 4-7: 0.5 mg twice daily; Days 8-14: 1 mg twice daily. This will appear identical to the drug Varenicline, but will be a placebo.

SUMMARY:
The objective is to provide a preliminary test of the ability of two pharmacological treatments, the nicotine nasal spray and varenicline, relative to placebos, to reduce smoking during the 4 hours following methadone dosing.

DETAILED DESCRIPTION:
Smoking prevalence is over 83% in methadone-maintained patients. These patients experience significant difficulty quitting, and there is evidence that a majority of methadone-maintained patients smoke most of their cigarettes in the 4 hours following methadone dosing. The objective is to provide a preliminary test of the ability of two pharmacological treatments, the nicotine nasal spray and varenicline, relative to placebos, to reduce smoking during the 4 hours following methadone dosing.

ELIGIBILITY:
Inclusion Criteria:

1. be male or female, 18 years of age or older
2. be able to understand the study, and having understood, provide written informed consent in English
3. have been enrolled in the University of Cincinnati Physicians Company-Opioid Treatment Program (UCPC-OTP) program for at least 30 days and be stable on the current methadone dose for at least 1 week
4. have smoked cigarettes for at least 3 months, have a measured exhaled carbon monoxide (CO) level > 8 parts per million (ppm), and not planning to seek smoking-cessation treatment within the next 3 months
5. have a willingness to comply with all study procedures, including trying to stop smoking during designated weeks, and to comply with medication instructions
6. based on a week of Quitbit cigarette lighter assessments, with at least 5 days of usable data, smoke ≥ 10 cigarettes/day and smoke at least 30% of daily cigarettes within the 4-hour post-methadone-dosing period
7. if female and of child bearing potential, agree to use one of the following methods of birth control: oral contraceptives, contraceptive patch, barrier (diaphragm or condom), intrauterine contraceptive system, levonorgestrel implant, medroxyprogesterone acetate contraceptive injection,complete abstinence from sexual intercourse, hormonal vaginal contraceptive ring.

Exclusion Criteria:

1. have a current or past diagnosis of any psychotic disorder, or bipolar I or II disorder
2. have a psychiatric condition that, in the judgment of the study physician would make study participation unsafe or which would make treatment compliance difficult
3. be a significant suicidal/homicidal risk
4. have a medical condition that, in the judgment of the study physician, would make study participation unsafe or which would make treatment compliance difficult. Such conditions include, but are not limited to:

   * liver function tests greater than 3 times upper limit of normal
   * serum creatinine greater than 2 mg/dL
5. have had clinically significant cardiovascular or cerebrovascular disease within the past 6 months or have clinically significant ECG abnormalities
6. have taken an investigational drug within 30 days before consent
7. be taking concomitant medications that are contraindicated for use with the NNS or varenicline
8. be taking any concomitant medications that could increase the likelihood of smoking cessation (such as wellbutrin or nortriptyline)
9. have a known or suspected hypersensitivity to varenicline or the nicotine nasal spray (NNS)
10. use/have used smoking-cessation counseling programs with individual counseling or smoking-cessation medication treatments currently, or within 30 days before consent
11. have used electronic cigarettes or tobacco products, other than cigarettes, in the week before consent
12. be pregnant or breastfeeding
13. be anyone who, in the judgment of the investigator, would not be expected to complete the study protocol (e.g., due to relocation from the clinic area, probable incarceration, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2016-03; Primary Completion 2017-08-25 (Actual); Study Completion 2017-08-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theresa Winhusen, PhD, Principal Investigator — University of Cincinnati
Locations (1):
- UC Physicians Company, LLC Opioid Treatment Program, Cincinnati, Ohio, United States

REFERENCES:
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Order 1 | Order 2 | Order 3 | Order 4
Started | 2 | 2 | 1 | 2
Completed | 1 | 2 | 1 | 2
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants randomized in this crossover trial (each randomized participant was intended to receive each medication)
Arm/Group | All Participants
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.9 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race, Ethnicity: White, Non-Hispanic | 6
  Race, Ethnicity: Other, Non-Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 7
Fagerström Test for Nicotine Dependence [Mean (Standard Deviation); unit: units on a scale] — Scores can range from a minimum of 0 to a maximum of 10. Higher scores represent more severe nicotine dependence.
  units on a scale | 5.3 (1.0)
Years in Methadone Treatment [Mean (Standard Deviation); unit: years] | 3.1 (3.6)
Current Methadone Dose [Mean (Standard Deviation); unit: milligrams] | 109.9 (35.0)

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Daily Cigarettes Smoked in the 4 Hours After Receiving Methadone Dose
Description: Subjects will be given a special electronic cigarette lighter called Quitbit.The electronic lighter will record a timestamp for each time the lighter is used to light a cigarette. Data will be collected from the lighter at each study visit. This will measure how many cigarettes are smoked and when.
Time Frame: 7 weeks
Population: Varenicline and placebo varenicline analysis populations are less than 7 because 1 participant was lost to follow-up and provided no data for these assigned medications.
Measure: Mean (Standard Deviation); unit: proportion of daily cigarettes
Groups:
- Nicotine Nasal Spray: All participants who received the nicotine nasal spray
- Placebo Nasal Spray: All participants who received the placebo nasal spray
- Varenicline Tablets: All participants who received the active varenicline tablets
- Placebo Varenicline Tablets: All participants who received the placebo varenicline tablets
Arm/Group | Nicotine Nasal Spray | Placebo Nasal Spray | Varenicline Tablets | Placebo Varenicline Tablets
Number analyzed (Participants) | 7 | 7 | 6 | 6
proportion of daily cigarettes | 0.294 (0.130) | 0.177 (0.104) | 0.196 (0.088) | 0.325 (0.346)

2. Secondary Outcome: Cigarettes Per Day
Description: The Quitbit lighter will measure how many cigarettes are smoked per day. In addition to the Quitbit lighter measurement, the Timeline Follow Back (TLFB) form will be filled out for each subject to measure use, as well.
Time Frame: 7 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cigarettes per day
Arm/Group | Nicotine Nasal Spray | Placebo Nasal Spray | Varenicline Tablets | Placebo Varenicline Tablets
Number analyzed (Participants) | 7 | 7 | 6 | 6
cigarettes per day | 13.7 (6.4) | 15.8 (8.2) | 12.5 (12.8) | 9.0 (6.9)

3. Secondary Outcome: Number of Participants With Carbon Monoxide Levels Less Than or Equal to 8 Parts-per-million
Description: Carbon monoxide (CO) in each participant's breath will be tested. A CO level less than or equal to 8 parts-per-million will be used to verify reports of no smoking.
Time Frame: up to 8 weeks
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nicotine Nasal Spray | Placebo Nasal Spray | Varenicline Tablets | Placebo Varenicline Tablets
Number analyzed (Participants) | 7 | 7 | 6 | 6
Participants
  Participants with CO less than or equal to 8 ppm | 2 | 1 | 3 | 2
  Participants with CO greater than 8 ppm | 5 | 6 | 3 | 4

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Nicotine Nasal Spray | Placebo Nasal Spray | Varenicline Tablets | Placebo Varenicline Tablets
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 4/7 | 1/7 | 2/6 | 0/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Nicotine Nasal Spray (N=7) | Placebo Nasal Spray (N=7) | Varenicline Tablets (N=6) | Placebo Varenicline Tablets (N=6)
sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ear ache (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
headache (Nervous system disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
flu-like symptoms (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
hot / cold flashes (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
difficulty hearing in right ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
bloodshot eyes (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
menstrual cramps (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-17): https://cdn.clinicaltrials.gov/large-docs/32/NCT02147132/Prot_SAP_000.pdf